CLINICAL TRIAL: NCT03592316
Title: Impact of a Lower Extremity Amputation Pathway Protocol in Dysvascular Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018021
Record Dates: First submitted 2018-07-10; First posted 2018-07-19 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Lower Extremity Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lower Extremity Amputation Pathway (Experimental): Patients will follow the Lower Extremity Amputation Pathway, which will include pre-operative consultations and earlier progression with physical therapy post-operatively.
  Interventions: Other: Lower Extremity Amputation Pathway

INTERVENTIONS:
Other: Lower Extremity Amputation Pathway — Pre-operatively: Subjects will meet with social work/case management, physical therapy, anesthesiology, and the prosthetist for the following: discuss expectations and rehabilitation; pain control options and consideration for epidural or nerve block; prosthetic treatment and care timeline.
  Post-operatively: Physical therapy will begin on post-op day 1 with increasing complexity through post-op day 3. On post-op day 3 the wound will be examined by the surgeon and subjects will be cleared for discharge.
  Quality of life surveys will be given at several time points during post-operative care.

SUMMARY:
The LEAP protocol is a prospective cohort study of dysvascular patients designed to determine whether implementation of a multi-disciplinary lower extremity amputation protocol in the peri-operative period can shorten post-operative length of stay in patients undergoing trans-tibial or trans-femoral amputations. A consecutive sample of patients diagnosed with peripheral vascular disease and/or diabetes requiring major lower extremity amputation will be enrolled in the study and compared to retrospective controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age diagnosed with peripheral vascular disease and/or diabetes mellitus
* Patients undergoing trans-tibial or trans-femoral amputations

Exclusion Criteria:

* Patients undergoing amputation for trauma, malignancy, or necrotizing fasciitis with no dysvascular diagnosis
* Patients who have previously undergone an amputation
* Patients who were unable to function independently prior to admission
* Patients admitted to the ICU prior to surgery
* Attending surgeon does not approve of the patient being enrolled
* Prisoners
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | Through hospital discharge, approximately 3 days after surgery
  The total hospital length of stay for the lower extremity amputation admission

SECONDARY OUTCOMES:
Mortality | Up to 6 months after surgery
  Mortality during the follow-up period
Major adverse limb event | Up to 6 months after surgery
  Hematoma, infection, ischemia, and/or need for revision of amputation
In-hospital morbidity | Through hospital discharge, approximately 3 days after surgery
  Catheter Associated Urinary Tract Infection, Pneumonia, Deep Vein Thrmbosis, and/or Pulmonary Embolism
Return to functional independence | Up to 6 months after surgery
  Time to return to functional independence at home

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Ann O'Banion, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Community Regional Medical Center, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No